CLINICAL TRIAL: NCT02947568
Title: Genetical Background of Non-alcoholic Fatty Liver Disease (NAFLD) in Diabetes Mellitus and in Chronic Kidney Disease
Acronym: NAFLDDMCKD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Pecs (Other)
Collaborators: Teaching Hospital Markusovszky, Szombathely (Unknown); Fresenius Medical Care North America (Industry)
Responsible Party: Principal Investigator, Dr. Gergő Molnár, MD, University of Pecs
Other Study IDs: Pecs_NAFLD_01
Record Dates: First submitted 2016-09-22; First posted 2016-10-28 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Non-alcoholic Fatty Liver Disease; Chronic Kidney Disease; Diabetes Mellitus
Keywords: Non-alcoholic Fatty Liver Disease; Chronic Kidney Disease; Diabetes Mellitus; Cross-sectional
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Renal Insufficiency, Chronic; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CKD: chronic kidney disease
  Interventions: Other: non-interventional study
- DM: diabetes mellitus
  Interventions: Other: non-interventional study
- CKD+DM: chronic kidney disease + diabetes mellitus
  Interventions: Other: non-interventional study

INTERVENTIONS:
Other: non-interventional study

SUMMARY:
The present study investigates relationship between non-alcoholic fatty liver disease and its risk factors, such as genetic background and diseases, such as chronic kidney disease and diabetes mellitus.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is a multisystemic disease, also affecting extrahepatic organs (1,2,6). According to former data, not only the prevalence of chronic hepatic disease, chronic cardiovascular diseases, but also the prevalence of chronic kidney disease (CKD) is higher in NAFLD (4,7). A strong association has been shown between diabetes mellitus (DM) and NAFLD as well (3,5,10).

Many genetical factors have been studied in the background of NAFLD. Many studies have proved the effect of patatin-like phospholipase domain-containing protein 3 gene (PNPLA3) (8,9). Effect of numerous genetical polymorphisms has been suggested behind oxidative stress responsible for NAFLD (8).

ELIGIBILITY:
Inclusion Criteria:

* CKD (renal replacement therapy non excluded)
* DM
* CKD+DM

Exclusion Criteria:

* alcohol abuse

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CKD without DM, or patients with DM without CKD, or patients with both CKD and DM, aged 18-90
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Association of NFS (NAFLD fibrosis score) and HSI (hepatic steatosis index) with underlying conditions | 2 years
  The association of hepatic steatosis with chronic kidney disease, diabetes mellitus and the the persence of these two will be assessed
Association of genetical factors with NFS and HSI | 2 years
  The association of hepatic steatosis with genetic factors will be assessed. In case of patatin-like phospholipase domain-containing protein 3 gene (PNPLA3) : rs738409, rs2281135, rs2294918 single nuclear polimorfism (SNP) will be examined

SECONDARY OUTCOMES:
Association of hepatic steatosis with renal function | 2 years
  The association of serum creatinine, eGFR, blood urea nitrogen, serum sodium, serum potassium, serum calcium with NFS and HSI will be assessed
Association of glucose metabolism parameters with hepaic steatosis indices | 2 years
  Association of HbA1C, fructosamine, blood glucose, serum insulin, HOMAIR, serum uric acid with NFS and HSI
Association of liver function and hepatic setatosis indices | 2 years
  Association of serum bilirubine, serum GOT, serum GPT, serum GGT, serum ALP, serum LDH, INR, serum total protein, serum albumin with NFS and HSI
Association of serum lipid profile and hepatic setatosis indices | 2 years
  Association of serum total cholesterol, serum HDL-cholesterol, serum LDL-cholesterol, serum triglyceride, serum carnitine with NFS and HSI
Association of iron metabolism parameters with hepatic setatosis indices | 2 years
  association of serum iron, serum transferrine, serum transferrine saturation, serum ferritine with NFS and HSI
The relationship between blood count, sedimentation and inflammation with hepatic setatosis indices | 2 years
  Association of blood count, erythrocyte sedimentation rate, CRP with NFS and HSI
Assotion of serum proteins with hepatic setatosis indices | 2 years
  association of urinary total protein, urinary albumin, urinary total protein/creatinine ratio, urinary albumin/creatinine ratio with NFS and HSI
Association of pathological tyrosine isoforms with hepatic setatosis indices | 2 years
  Association of serum meta-Tyr, serum ortho-Tyr, urinary meta-Tyr, urinary ortho-Tyr, urinary meta-Tyr/creatinine ratio, urinary ortho-Tyr/creatinine ratio with NFS and HSI

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Medicine and Nephrological Center, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Alp H, Karaarsian S, Selver EB,Atabek ME, Altin H, Baysal T. Association between nonalcoholic fatty liver disease and cardiovascular risk in obese children and adolescents. Can J Cardiol 2013;29:1118-1125. 2. Byrne CD, Targher G: NAFLD: A multisystem disease. Review. Journal of Hepatology, 2015; 62:S47-S64. 3. Kasturiratne A, Weerasinghe S, Dassanayake AS, rajindrajith S, de Silva AP, Kato N, et al. Influence of non-alcoholic fatty liver disease on the development of diabetes mellitus. J Gastroenterol Hepatol 2013;60:384-391. 4. Li G, Shi W, Hug H, Chen Y, Liu L, Yin D. Nonalcoholic fatty liver disease associated with impairment of kidney function in nondiabetes population. Biochem Med 2012;22:92-99. 5. Okamoto M, Takeda Y, Yoda Y, Kobayashi K, Fujino MA, Yamagata Z. The association of fatty liver and diabetes risk. J Epidemiol 2003;13:15-21. 6. Pacifico L, Di MM, De MA, Bezzi M, Osborn JF, Catalano C, et al. Left ventricular dysfunction in obese children and adolescents with nonalcoholic fatty liver disease. Hepatology 2014;59:461-470. 7. Targher G, Choncol MB, Byrne CD. CKD a nonalcoholic fatty liver disease. Am J Kidney Dis 2014;64:638-652. 8. Wood KL, Miller MH, Dillon JF. systematic review of genetic association studies involving histologically confirmed non-alcoholic fatty liver disease BMJ Open Gastro 2015:2:e000019. doi10.1136/bmjgast-2014-000019 9. Zain SM, Mohamed R, Hyogo H, et al. A multi-ethnic study of a PNPLA3 variant and its association with disease severity in non-alcoholic fatty liver disease. Hum genet 2012;131:1145-1152. 10. Zuppini G, Fedeli U, Gennaro N, Saugo M, Targher G, Bonora E. Mortality from chronic liver diseases in diabetes. Am J Gastroenterol 2014;109:1020-1025.